CLINICAL TRIAL: NCT04286841
Title: The Real World Study of Neoadjuvant Immunotherapy in Early Stage NSCLC in China
Status: Recruiting | Type: Observational
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: RW1804
Record Dates: First submitted 2019-10-16; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Immunotherapy; Lung Cancer
Keywords: neoadjuvant immunotherapy; NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant immunotherapy
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Patients in this group should be histologically confirmed potentially resectable NSCLC with stage II-IIIA. Furthermore patients would receive either single agent immunotherapy or immunotherapy combined with chemotherapy.

SUMMARY:
Several published clinical trials have shown the superiority of immunotherapy in neoadjuvant setting. Here we conducted this real world study to see whether neoadjuvant immunotherapy would bring MPR and survival benefits in NSCLC, for example, single agent immunotherapy or immunotherapy combination with chemotherapy. Furthermore biomarker analysis would be also performed to achieve personalized neoadjuvant immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided
* Males or females aged ≥18 years
* Able to comply with the required protocol and follow-up procedures、
* Pathologically diagnosed of potentially resectable non-small cell lung cancer with stage II-IIIA (TNM 8th edition)
* Measurable disease must be characterized according to RECIST 1.1 criteria
* ECOG performance status 0-1
* Regardless of PD-L1 expression
* EGFR mutation (-) and ALK translocation (-)
* Pulmonary function could be well tolerated by lobectomy or pneumonectomy

Exclusion Criteria:

* EGFR mutation (+) or ALK translocation (+)
* Active Central nervous system (CNS) metastases
* Patients with active, known or suspected autoimmune disease.
* Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement or unexpected conditions of recurrence in the absence of an external trigger are allowed to be included
* Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment
* Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Patients with a history of interstitial lung disease cannot be included if they have symptomatic ILD (Grade 3-4) and/or poor lung function. Patients with other active malignancy requiring concurrent intervention and/ or concurrent treatment with other investigational drugs or anti-cancer therapy
* Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/ dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period
* Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information
* Patients who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways Patients with positive test for hepatitis B virus surface antigen (HBVsAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating active hepatitis
* Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) Patients with history of allergy to study drug components excipients
* Women who are pregnant or in the period of breastfeeding
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study
* In case of doubt please contact trial team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IIA-IIIA NSCLC
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
MPR | From the date of surgery up to 10 weeks
  To evaluate the major pathological response (MPR) rate of participants

SECONDARY OUTCOMES:
Objective Response Rate | From the date of surgery up to 10 weeks
  Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
MPR based on diverse PD-L1 expression | From the date of surgery up to 10 weeks
  Percentage of Participants with Major Pathologic Response Rates For Programmed Death Ligand 1 (PD-L1)-Positive Versus PD-L1-Negative Participants
Percentage of Participants with Adverse Events | From the date of the first cycle of neoadjuvant treatment until 90 days after end of treatment, assessed up to 100 months
  No delayed resection rate and incidence of adverse event (AE)/serious adverse event (SAE)
Progression Free Survival (PFS) | From date of the first cycle of neoadjuvant treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression Free Survival

OTHER OUTCOMES:
Pathological Complete Response (pCR) | From the date of surgery up to 10 weeks
  Evaluation of the pathological complete response: The pathological complete response is defined as the absence of residual tumor in lung and lymph nodes in patients treated with chemo-immunotherapy versus patients treated with chemotherapy alone

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided